CLINICAL TRIAL: NCT05785741
Title: A Phase 1/2a, Multicenter, Open-Label, First in Human Study to Assess the Safety, Tolerability, Pharmacokinetics, and Preliminary Antitumor Activity of DB-1310 in Subjects With Advanced/Metastatic Solid Tumors
Brief Title: A Study of DB-1310 in Advanced/Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: DualityBio Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DB-1310-O-1001; CTR20231736 (Other: CENTER FOR DRUG EVALUATION, NMPA)
Record Dates: First submitted 2023-03-14; First posted 2023-03-27 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Advanced Solid Tumor
Keywords: HER3; NSCLC; CRPC; HNSCC; BC; non-small cell lung cancer; castration-resistant prostate cancer; head and neck squamous cell carcinoma; breast cancer; ESCC; BTC
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Carcinoma, Non-Small-Cell Lung; Breast Neoplasms | interventions — Trastuzumab; osimertinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (24):
- DB-1310 Dose Level 1 (Experimental): Enrolled Subjects will receive a single-dose of DB-1310 at Dose Level 1 on Day 1 of each cycle Q3W
  Interventions: Drug: DB-1310
- DB-1310 Dose Level 2 (Experimental): Enrolled Subjects will receive a single-dose of DB-1310 at Dose Level 2 on Day 1 of each cycle Q3W
  Interventions: Drug: DB-1310
- DB-1310 Dose Level 3 (Experimental): Enrolled Subjects will receive a single-dose of DB-1310 at Dose Level 3 on Day 1 of each cycle Q3W
  Interventions: Drug: DB-1310
- DB-1310 Dose Level 4 (Experimental): Enrolled Subjects will receive a single-dose of DB-1310 at Dose Level 4 on Day 1 of each cycle Q3W
  Interventions: Drug: DB-1310
- DB-1310 Dose Level 5 (Experimental): Enrolled Subjects will receive a single-dose of DB-1310 at Dose Level 5 on Day 1 of each cycle Q3W
  Interventions: Drug: DB-1310
- DB-1310 Dose Level 6 (Experimental): Enrolled Subjects will receive a single-dose of DB-1310 at Dose Level 1 on Day 1 of each cycle Q3W
  Interventions: Drug: DB-1310
- DB-1310 Dose Level 7 (Experimental): Enrolled Subjects will receive a single-dose of DB-1310 at Dose Level 1 on Day 1 of each cycle Q3W
  Interventions: Drug: DB-1310
- DB-1310 Dose Level 8 (Experimental): Enrolled subjects with HER2 positive BC who will receive DB-1310 on a selected dose level in combination with Trastuzumab
  Interventions: Drug: DB-1310; Drug: Trastuzumab
- DB-1310 Dose Level 9 (Experimental): Enrolled subjects with HER2 positive BC who will receive DB-1310 on a selected dose level in combination with Trastuzumab
  Interventions: Drug: DB-1310; Drug: Trastuzumab
- DB-1310 Dose Level 10 (Experimental): Enrolled subjects with HER2 positive BC who will receive DB-1310 on a selected dose level in combination with Trastuzumab
  Interventions: Drug: DB-1310; Drug: Trastuzumab
- DB-1310 Dose Level 11 (Experimental): Enrolled subjects with NSCLC subjects with EGFR Ex19del or L858R, G719X, S768I, L861Q alone or in combination with other EGFRm who will receive DB-1310 on a selected dose level in combination with Osimertinib
  Interventions: Drug: DB-1310; Drug: Osimertinib
- DB-1310 Dose Level 12 (Experimental): Enrolled subjects with NSCLC subjects with EGFR Ex19del or L858R, G719X, S768I, L861Q alone or in combination with other EGFRm who will receive DB-1310 on a selected dose level in combination with Osimertinib
  Interventions: Drug: DB-1310; Drug: Osimertinib
- DB-1310 Dose Level 13 (Experimental): Enrolled subjects with NSCLC subjects with EGFR Ex19del or L858R, G719X, S768I, L861Q alone or in combination with other EGFRm who will receive DB-1310 on a selected dose level in combination with Osimertinib
  Interventions: Drug: DB-1310; Drug: Osimertinib
- DB-1310 Dose Expansion 1 (Experimental): Enrolled Subjects with advanced/unresectable, or metastatic adenocarcinoma NSCLC with EGFR activating mutation who have progressed on or after standard systemic treatments will receive a single-dose of DB-1310 on a selected dose level (RP2D) Day 1 of each cycle Q3W
  Interventions: Drug: DB-1310
- DB-1310 Dose Expansion 2 (Experimental): Enrolled Subjects with advanced/unresectable, or metastatic NSCLC without EGFR activating mutation who have progressed on or after standard systemic treatments will receive a single-dose of DB-1310 on a selected dose level (RP2D) Day 1 of each cycle Q3W
  Interventions: Drug: DB-1310
- DB-1310 Dose Expansion 3 (Experimental): Enrolled Subjects with advanced/unresectable, or metastatic CRPC who have progressed on or after standard systemic treatments will receive a single-dose of DB-1310 on a selected dose level (RP2D) Day 1 of each cycle Q3W
  Interventions: Drug: DB-1310
- DB-1310 Dose Expansion 4 (Experimental): Enrolled Subjects with advanced/unresectable, or metastatic HNSCC who have progressed on or after standard systemic treatments will receive a single-dose of DB-1310 on a selected dose level (RP2D) Day 1 of each cycle Q3W
  Interventions: Drug: DB-1310
- DB-1310 Dose Expansion 5 (Experimental): Enrolled Subjects with advanced/unresectable, or metastatic BC with HER2-positive (IHC3+, or IHC2+ and ISH+) who have progressed on or after HER2 targeted systemic treatments will receive a single-dose of DB-1310 on a selected dose level Day 1 of each cycle Q3W in combination with trastuzumab deruxtecan.
  Interventions: Drug: DB-1310; Drug: Trastuzumab
- DB-1310 Dose Expansion 6 (Experimental): Enrolled Subject with other advanced/unresectable, or metastatic solid tumors who have progressed on or after standard systemic treatment, or for which no standard systemic treatment is available will receive a single-dose of DB-1310 on a selected dose level (RP2D) Day 1 of each cycle Q3W
  Interventions: Drug: DB-1310
- DB-1310 Dose Expansion 7 (Experimental): Enrolled subjects with advanced/unresectable, or metastatic non-squamous NSCLC with EGFR exon 19 deletion or L858R mutation who haven't received any treatment in locally advanced, or metastatic disease will receive a single-dose of DB-1310 on a selected dose level Day 1 of each cycle Q3W in combination with Osimertinib.
  Interventions: Drug: DB-1310; Drug: Osimertinib
- DB-1310 Dose Expansion 8 (Experimental): Enrolled subjects with NSCLC with EGFR who will receive DB-1310 on a selected dose level in combination with Osimertinib
  Interventions: Drug: DB-1310; Drug: Osimertinib
- DB-1310 Dose Expansion 9 (Experimental): Enrolled subjects with NSCLC with KRAS mutation who will receive DB-1310 on a selected dose level (RP2D)
  Interventions: Drug: DB-1310
- DB-1310 Dose Expansion 10 (Experimental): Enrolled subjects with ESCC who will receive DB-1310 on a selected dose level (RP2D)
  Interventions: Drug: DB-1310
- DB-1310 Dose Expansion 11 (Experimental): Enrolled subjects with BTC who will receive DB-1310 on a selected dose level (RP2D)
  Interventions: Drug: DB-1310

INTERVENTIONS:
Drug: DB-1310 — Administered I.V.
Drug: Trastuzumab — Administered I.V.
  Arms: DB-1310 Dose Expansion 5; DB-1310 Dose Level 10; DB-1310 Dose Level 8; DB-1310 Dose Level 9
Drug: Osimertinib — Oral
  Arms: DB-1310 Dose Expansion 7; DB-1310 Dose Expansion 8; DB-1310 Dose Level 11; DB-1310 Dose Level 12; DB-1310 Dose Level 13

SUMMARY:
This is a dose-escalation and dose-expansion Phase 1/2a trial to evaluate the safety and tolerability of DB-1310 in subjects with advanced solid tumors.

DETAILED DESCRIPTION:
This is a multicenter, open-label, multiple-dose, FIH Phase 1/2a study. Phase 1 adopts the standard "3+3" design to identify: the MTD and/or RP2D of DB-1310 as monotherapy, the RCD_A of DB-1310 in combination with trastuzumab or approved trastuzumab biosimilar and the RCD_B of DB-1310 in combination with Osimertinib; Phase 2a is a dose expansion phase to confirm the safety, tolerability and explore efficacy in selected malignant solid tumors treated with DB-1310 as monotherapy or in combination with trastuzumab or approved trastuzumab biosimilar or in combination with Osimertinib.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female adults (defined as ≥ 18 years of age or acceptable age according to local regulations at the time of voluntarily signing of informed consent).
2. Have relapsed or progressed on or after standard systemic treatments, or intolerable with standard treatment, or for which no standard treatment is available. Documented radiological disease progression during/after most recent treatment regimen for advanced/unresectable, or metastatic disease.
3. At least one measurable lesion as assessed by the investigator according to response evaluation criteria in solid tumors (RECIST) version 1.1 criteria.
4. Has a life expectancy of ≥ 3 months.
5. Has an Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0-1.
6. Has LVEF ≥ 50% by either echocardiography (ECHO) or multiple-gated acquisition (MUGA) within 28 days before enrollment.
7. Has adequate organ functions within 7 days prior to Day 1 of Cycle 1.
8. Has adequate treatment washout period prior to Day 1 of Cycle 1.
9. Is willing to provide pre-existing resected tumor samples or undergo fresh tumor biopsy for the measurement of HER3 level and other biomarkers if no contraindication. For HER2 IHC 0 breast cancer subjects, it is highly recommended to collect additional tumor sample (Refer to Lab Manual).
10. Is capable of comprehending study procedures and risks outlined in the informed consent and able to provide written consent and agree to comply with the requirements of the study and the schedule of assessments.
11. Male and female subjects of reproductive/childbearing potential must agree to use adequate contraceptive methods (e.g., double barrier or intrauterine contraceptive) during the study and for at least 4 months and 7 months after the last dose of study drug, respectively.

    Females must be using highly effective contraceptive measures during the study and for at least 7 months after the last dosing of study drug, and must have a negative pregnancy test prior to start of dosing if of child-bearing potential, or must have evidence of non-child-bearing potential by fulfilling one of the following criteria at screening:
    * Post-menopausal defined as aged 50 years or more and amenorrhoeic for at least 12 months following cessation of all exogenous hormonal treatments
    * Women under 50 years old would be considered postmenopausal if they have been amenorrhoeic for 12 months or more following cessation of exogenous hormonal treatments and with LH and FSH levels in the post-menopausal range for the institution
    * Documentation of irreversible surgical sterilization by hysterectomy, bilateral oophorectomy or bilateral salpingectomy but not tubal ligation
12. Male subjects must not freeze or donate sperm starting at screening and throughout the study period, and at least 4 months after the final study drug administration.
13. Female subjects must not donate, or retrieve for their own use, ova from the time of screening and throughout the study treatment period, and for at least 7 months after the final study drug administration.

Exclusion Criteria:

1. Prior treatment with HER3 targeted therapy.
2. Prior treatment with antibody drug conjugate with topoisomerase I inhibitor (except trastuzumab deruxtecantopoisomerase I inhibitor HER2 ADC for backfilled subjects in Combo A of Phase 1 and subjects in Cohort 2e of Phase 2a, and not applicable for subjects enrolled for DLT observation in Phase 1).
3. Has a medical history of symptomatic congestive heart failure (CHF) (New York Heart Association [NYHA] classes II-IV) or serious cardiac arrhythmia requiring treatment.
4. Has a medical history of myocardial infarction or unstable angina within 6 months before enrollment.
5. Has any clinically important abnormalities in rhythm, conduction or morphology of resting electrocardiogram (ECG), e.g., complete left bundle branch block, third-degree heart block, second-degree heart block, or PR interval > 250 milliseconds (ms).
6. Has an average of Fredericia's formula-QT corrected interval (QTcF) prolongation to > 470 millisecond (ms) in males and females based on a 12-lead electrocardiogram (ECG) in triplicate.
7. Unable or unwilling to discontinue concomitant drugs that are known to prolong the QT interval.

   For Combo B of Phase 1 and Cohort 2g, 2k of Phase 2a, patients currently receiving (or unable to stop use prior to receiving the first dose of Osimertinib) medications or herbal supplements known to be strong inducers of CYP3A4 (at least 3-week prior) (refer to Section 6.9.1) are ineligible, and all patients must try to avoid concomitant use of any medications, herbal supplements and/or ingestion of foods with known inducer effects on CYP3A4.
8. Has a history of (non-infectious) ILD/pneumonitis and/or radiation pneumonitis that required steroids, has current ILD/pneumonitis and/or radiation pneumonitis, or where suspected ILD/pneumonitis and/or radiation pneumonitis cannot be ruled out by imaging at screening.
9. Have a lung-specific intercurrent clinically significant illness including, but not limited to, any underlying pulmonary disorder (e.g., pulmonary emboli within 3 months prior to Cycle 1 Day 1, severe asthma, severe chronic obstructive pulmonary disorder, restrictive lung disease, significant pleural effusion etc.), and any autoimmune, connective tissue or inflammatory disorder with pulmonary involvement (e.g., rheumatoid arthritis, Sjogren's syndrome, sarcoidosis etc.), and/or prior pneumonectomy (complete).
10. Has an uncontrolled infection requiring intravenous injection of antibiotics, antivirals, or antifungals.
11. Has clinically significant corneal disease.
12. Know human immunodeficiency virus (HIV) infection.
13. Subjects have active viral (any etiology) hepatitis are excluded. However, subjects with positive hepatitis B surface antigen (HBsAg) who have the HBV DNA (viral load) below the lower limit quantification or HBV DNA titer < 1000 cps/mL or 100 IU/mL per local testing and are not currently on viral suppressive therapy may be eligible and should be discussed with the Sponsor's Medical Monitor. However, subjects with a history of hepatitis C virus (HCV) infection who have completed curative antiviral treatment and have the HCV RNA below the lower limit of quantification per local testing are eligible for study entry.
14. Is a lactating mother (women who are willing to temporarily interrupt breastfeeding will also be excluded), or pregnant as confirmed by serum pregnancy tests performed within 7 days prior to Cycle 1 Day 1.
15. Has clinically active brain metastases, defined as untreated and symptomatic, or requiring therapy with steroids or anticonvulsants to control associated symptoms. However, subjects with asymptomatic central nervous system (CNS) metastases who are radiologically and neurologically stable for at least 4 weeks following CNS-directed therapy, and who are on stable or decreasing doses of corticosteroids equivalent to ≤10 mg/day prednisone are eligible for study entry.
16. Has unresolved toxicities from previous anticancer therapy, defined as toxicities (other than alopecia) not yet resolved to NCI-CTCAE version 5.0, grade ≤ 1 or baseline. Subjects with chronic Grade 2 toxicities (e.g., Grade 2 neuropathy) may be eligible based on the discussion and agreement between Investigator and Sponsor.
17. Has multiple primary malignancies within 3 years before enrollment, except adequately resected non-melanoma skin cancer (e.g., resected basal or squamous cell skin cancer), curatively treated in-situ disease (e.g., carcinoma in situ of the cervix or breast), other solid tumors curatively treated (e.g., superficial bladder cancer), or contralateral breast cancer.
18. Has substance abuse or any other medical conditions that would increase the safety risk to the subject or interfere with participation or evaluation of the clinical study in the opinion of the investigator.
19. Has known hypersensitivity to either the drug substances or inactive ingredients in the drug product.
20. Patients with other reasons that, in the opinion of the Investigator, make them unsuitable to participate in this study.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2023-04-10 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Percentage of Participants with Dose-Limiting Toxicities (DLTs) as assessed by CTCAE v5.0. Percentage of participants in Part 1 with DLTs | up to 21 days after Cycle 1 Day 1
  Percentage of participants in Part 1 with DLTs
Phase 1: Percentage of Participants with Treatment Emergent Adverse Events (TEAEs) as assessed by CTCAE v5.0. | Up to follow-up period, approximately 1 year post-treatment
  Percentage of participants with TEAE in Part 1 graded according to NCI CTCAE v5.0
Phase 1: Percentage of Participants with Serious Adverse Events (SAEs) as assessed by CTCAE v5.0. | Up to follow-up period, approximately 1 year post-treatment
  Percentage of Participants with SAEs in Part 1 graded according to NCI CTCAE v5.0
Maximum Tolerated Dose (MTD) of DB-1310 | 12 months
  MTD on the data collected during Part 1
Phase 1: Recommended Phase 2 Dose (RP2D) of DB-1310 | 12 months
  RP2D of DB-1310 based on the data collected during Part 1
Phase 2a: Percentage of Participants with Treatment Emergent adverse events (TEAEs) as assessed by CTCAE v5.0. | Up to follow-up period, approximately 1 year post-treatment
  Percentage of participants with TEAE in Part 2 graded according to NCI CTCAE v5.0
Phase 2a: Percentage participants with Serious Adverse Events (SAEs) as assessed by CTCAE v5.0. | Up to follow-up period, approximately 1 year post-treatment
  Percentage of participants with SAEs in Part 2 graded according to NCI CTCAE v5.0
Phase 2a: Percentage of Objective Response Rate (ORR) as assessed by RECIST 1.1. | Up to follow-up period, approximately 1 year post-treatment
  The percentage of subjects who had a best response rating of CR and PR, for Part 2 only which was maintained ≥4 weeks

SECONDARY OUTCOMES:
Phase 1 & Phase 2a: Pharmacokinetic-AUC | within 8 cycles (each cycle is 21 days)
  Area under the concentration-time curve from time 0 to infinity of DB-1310, total antibody and payload
Phase 1 & Phase 2a: Pharmacokinetic-Cmax | within 8 cycles (each cycle is 21 days)
  Maximum observed plasma concentration (Cmax) of DB-1310, total antibody and payload
Phase 1 & Phase 2a: Pharmacokinetic-Tmax | within 8 cycles (each cycle is 21 days)
  Time to Cmax of DB-1310, total antibody and payload
Phase 1 & Phase 2a: Pharmacokinetic-T1/2 | within 8 cycles (each cycle is 21 days)
  Phase 1 & Phase 2a: Pharmacokinetic-T1/2 of DB-1310, total antibody and payload
Phase 1: ORR will be determined from tumor assessments by investigator per RECIST 1.1 | with 8 cycles (each cycle is 21 days)
  Phase 1: ORR will be determined from tumor assessments by investigator per RECIST 1.1
Phase 1 & Phase 2a: duration of response (DoR) will be determined from tumor assessments by investigator per RECIST 1.1 | with 8 cycles (each cycle is 21 days)
  Phase 1 & Phase 2a: duration of response (DoR) will be determined from tumor assessments by investigator (by BICR in cohort 3 in Phase 2a) per RECIST 1.1
Phase 1 & Phase 2a: disease-control rate (DCR) | with 8 cycles (each cycle is 21 days)
  Phase 1 & Phase 2a: disease-control rate (DCR)
Phase 1 & Phase 2a: progression free survival (PFS) will be determined from tumor assessments by investigator per RECIST 1.1 | with 8 cycles (each cycle is 21 days)
  Phase 1 & Phase 2a: progression free survival (PFS) will be determined from tumor assessments by investigator per RECIST 1.1
Phase 1 & Phase 2a: overall survival (OS) | with 8 cycles (each cycle is 21 days)
  Phase 1 & Phase 2a: overall survival (OS)

CONTACTS AND LOCATIONS:
Overall Officials: Lily Hu, Study Director — DualityBio Inc.
Locations (21):
- United States (13):
  - University of California, Davis Comprehensive Cancer Center, Sacramento, California
  - UCLA Hematology/Oncology - Santa Monica, Santa Monica, California
  - D&H Cancer Research Center LLC, Margate, Florida
  - Sarah Cannon Research Institute at Florida Cancer Specialists, Orlando, Florida
  - BRCR global, Plantation, Florida
  - Florida Cancer Specialists, Sarasota, Florida
  - BRCR Medical Center Inc., Tamarac, Florida
  - Research Site 111, Atlanta, Georgia
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Carl & Edyth Lindner Center for Research & Education at The Christ Hospital and The Christ Hospital Cancer Center, Cincinnati, Ohio
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - NEXT Virginia, Fairfax, Virginia
- China (8):
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Hunan cancer hospital, Changsha, Hunan
  - Jiangsu Province hospital, Nanjing, Jiangsu
  - Affiliated Hospital of Jiangnan University, Wuxi, Jiangsu
  - The first hospital of Jilin University, Changchun, Jilin
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: No